CLINICAL TRIAL: NCT02156882
Title: Maputo Tuberculosis Trial Unit- Project (MaTuTU- Project)
Brief Title: Establishment of a Clinical Trial Unit in Mavalane, Maputo, in Mozambique
Acronym: MaTuTU
Status: Completed | Type: Observational
Sponsor: Michael Hoelscher (Other)
Responsible Party: Sponsor-Investigator, Michael Hoelscher, Prof. Dr., Ludwig-Maximilians - University of Munich
Organization: Ludwig-Maximilians - University of Munich (Other)
Other Study IDs: MaTuTU-TB-01
Record Dates: First submitted 2014-06-04; First posted 2014-06-05 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Tuberculosis
Keywords: TB; Tuberculosis; MaTuTU - Maputo Tuberculosis Trial Unit; Clinical Trial Capacity Development
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Sputum, Urine, Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- TB patients and Tb suspects: Patients with confirmed tuberculosis who are treated by the National TB Programme

SUMMARY:
In this longitudinal study with a follow up time of at least 6 months, up to 300 tuberculosis (TB) patients or TB suspects will be screened for TB using the Xpert MTB/RIF assay along with standard smear microscopy after Ziehl-Neelsen staining at the TB health clinic located at Mavalane health center. Confirmed TB cases will be followed up during TB therapy until month six after treatment initiation in order to obtain clinical and microbiological data on treatment including treatment response. Apart from relevant research questions in the field of TB diagnostics and treatment, the main objective of this study will be the development of a clinical TB research site, including capacity development in clinical and laboratory based TB research methods, in Mavalane, Maputo.

DETAILED DESCRIPTION:
Main study objective:

To assess the feasibility to perform a TB clinical trial in Maputo, Mozambique, by screening, examining,enrollment, follow-up and data collection of TB patients sent for TB treatment as well as TB suspects who are sent for smear microscopy to the TB clinic at the Mavalane health center.

Screening of study patients:

After consenting, each study participant (with confirmed or suspected TB) will be screened for TB with smear microscopy after Ziehl-Neelsen staining and Xpert MTB/RIF assay. In patients with signs of extrapulmonary TB manifestation, specimen collection other than sputum are to be decided by the treating physician in the patient' s best interest, to establish TB diagnosis by using smear microscopy and/or Xpert MTB/RIF assay. Patients without a positive Xpert MTB/RIF-assay result will not continue in the study but will be referred to the National TB Program for further evaluation and treatment. In patients with a positive Xpert MTB/RIF result in any specimen anti TB treatment will be commenced according to the National Guidelines. All TB positive study participants will be followed up until 6 months after TB treatment initiation.

Study methods:

Follow up visits will occur at week 1, 2, 4, 8, 12, 17 and 26 after commencement of TB therapy. An optional visit will be performed in selected patients at week 52 in order to confirm cure of TB disease. At each study visit, a clinical investigation will be performed and a medical questionnaire will be completed for each participant. Further, sputum and urine samples will be collected for the evaluation of the new TB diagnostics. A chest x-ray will be performed and blood for HIV testing, CD4 count, biochemistry and full blood picture will be collected at baseline only or when medically indicated during the course of the study.

Data recording and analysis:

The study will follow ethical principles as outlined in the declaration of Helsinki and its revisions (last in 2008) and will be performed in compliance with the guidelines of Good Clinical, Laboratory (GCLP) and Clinical Data Management Practice (GCDMP). All essential documents will be archived for 3 years. All patient information will be treated in a strictly confidential manner and will be linked to a unique ID number and not to personal identifiers. Data will be collected on paper CRFs, which will be entered into a secured clinical data management system, for which daily backups will be done. Double data entry will minimize data entry errors, and full data validation and cleaning process will be employed.

ELIGIBILITY:
Inclusion Criteria:

* >/= 18 years old
* Able and willing to give informed consent to study participation, including HIV-testing
* Positive TB result by Xpert MTB/RIF performed at the study clinic

Exclusion Criteria:

* TB treatment in the last 6 months
* Abandoned TB treatment at any time point in the past
* Suffering from a condition likely to lead to uncooperative behaviour e.g. psychiatric illness or alcoholism.
* Karnofsky index below 50%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: TB patients and TB suspects who present themselves or are referred to theTB clinic at the Mavalane Health center
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2014-06; Primary Completion 2016-05 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Number of participants with clinical and microbiological cure at month 6 after treatment initiation | 52 weeks in those patients which were enrolled until December 2014

CONTACTS AND LOCATIONS:
Overall Officials: Nilesh Bhatt, MD, MMED, Principal Investigator — Centro de Investigação e Treino em Saúde da Polana Caniço, Costa do Sol Street, nº 178, PO.BOX 264 Polana Caniço B neighborhood Maputo, Mozambique
Locations (2):
- Mozambique (2):
  - Centro de Investigação e Treino em Saúde da Polana Caniço, Maputo
  - Instituto Nacional de Saúde, Eduardo Mondlane Avenue nº 1008 MISAU, Maputo